CLINICAL TRIAL: NCT03941808
Title: Gastroprotected Superoxide Dismutase in Combination With UVB vs Placebo and UVB for Treating Vitiligo. A Randomized Double Blind Placebo Controlled Monocentric Study
Brief Title: Gastroprotected Superoxide Dismutase in Combination With UVB vs Placebo and UVB for Treating Vitiligo.
Acronym: Vitisod
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-PP-01
Record Dates: First submitted 2019-03-29; First posted 2019-05-08 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2020-10

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug (Experimental): 4 pills a day (1000mg) for 3 months then 2 pills a day (500 mg) for 3 months
  Interventions: Drug: Glisodin tablet
- Placebo (Placebo Comparator): 4 pills a day (1000mg) for 3 months then 2 pills a day (500 mg) for 3 months
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: Glisodin tablet — 4 pills a day (1000mg) for 3 months then 2 pills a day (500 mg) for 3 months
  Arms: Drug
Drug: Placebo tablet — 4 pills a day (1000mg) for 3 months then 2 pills a day (500 mg) for 3 months
  Arms: Placebo

SUMMARY:
The role of the oxidative stress in vitiligo is supported by many studies but robust data are lacking concerning their interest as therapeutic agents. The objective of the study is to compare the association of GLISODIN (a gastro-protected superoxide dismutase) and Nb-UVB to Nb-UVB and placebo for treating vitiligo.

Adult patients with non-segmental vitiligo affecting more than 5% of body surface area will be included.

The main criteria of evaluation will be the VES score at 6 months compared to baseline in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Vitiligo
* Vitiligo, SOD, UVB
* Non-segmental vitiligo with BSA>5%

Exclusion Criteria:

* Criteria of non-inclusion

  * Segmental or mixed vitiligo
  * Pregnancy
  * Vitiligo lesions localized only on hands and feet
  * Immuno-suppressive drugs
  * Corticosteroids
  * Photosensitive drugs
  * Photodermatosis
  * Personal history of skin cancer
  * Allergy to gluten

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-05-02 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Evaluation Vitiligo | At Baseline and at 6 weeks
  Change from Baseline VES (Vitiligo Extend Score) at 6 months

SECONDARY OUTCOMES:
Quality of life of patient | At Baseline and at 6 weeks
  Change from baseline DLQI at 6 months

OTHER OUTCOMES:
Vitiligo activity score | At baseline and at 6 months
  Change from vaseline SA-VES (self administrated VES) at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Passeron Thierry, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Passeron, Nice, Alpes-Maritime, France

IPD SHARING:
Plan to Share IPD: No